CLINICAL TRIAL: NCT07056361
Title: VOP/VIM Direct Electrical Stimulation Increases Motor Cortex Excitability and Motor Output
Brief Title: Stimulating Specific Brain Areas (VOP/VIM) With Electricity to Improve Movement and Muscle Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Gonzalez-Martinez (Other)
Responsible Party: Sponsor-Investigator, Jorge Gonzalez-Martinez, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY22100174
Record Dates: First submitted 2025-06-25; First posted 2025-07-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Movement Disorders (Incl Parkinsonism); Stroke; Traumatic Brain Injury; Brain Diseases; Parkinson Disease; Essential Tremor, Movement Disorders
MeSH Terms: conditions — Movement Disorders; Stroke; Brain Injuries, Traumatic; Brain Diseases; Parkinson Disease; Essential Tremor

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, open-label, descriptive, experimental.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Direct Cortical Stimulation and Deep Brain Stimulation of the Motor Thalamus (Experimental): Individuals undergoing deep brain stimulation device implanted in the motor thalamus for movement disorders treatment. Some of whom may also sustain speech, swallowing, and motor deficits.
  Interventions: Device: Direct cortical stimulation and deep brain stimulation of motor thalamus

INTERVENTIONS:
Device: Direct cortical stimulation and deep brain stimulation of motor thalamus — All participants enrolled will undergo implantation of deep brain stimulation electrode leads for treatment of movement disorders. In addition to standard-of-care subcortical mapping using micro-electrode recording (MER) and macrostimulation mapping during DBS placement, cortical local field potentials (LFPs) will be simultaneously recorded from primary motor (M1) and somatosensory (S1) cortical areas by placement of a temporary strip electrode (1X6) in the subdural space. The strip electrode over M1 will be used to produce motor evoked potentials to contralateral hand muscles from direct cortical stimulation (DCMEPs). Cortical and subcortical LFPs will be obtained alongside electromyographic (EMG) data while the patient performs contralateral upper extremity movement tasks and a variety of articulation exercises.

SUMMARY:
In this study the investigators aim to enroll patients scheduled to undergo deep brain stimulation (DBS) implantation for movement disorders for intra-operative testing. In addition to standard-of-care surgical procedure to implant deep brain stimulation electrode leads, participants will also be stimulated and recorded from cortical areas by a temporary strip electrode (1X6) in the subdural space. The electrodes will be connected to external stimulators and a series of experiments will be performed to assess effects of the DBS on movement quality and electrophysiology measures. Results of this study will elucidate the biological mechanisms related to deep brain stimulation in modulating motor and speech function in patients with abnormal movement disorders.

DETAILED DESCRIPTION:
In this study the investigators aim to enroll patients for intra-operative testing. Specifically, the investigators will recruit patients already undergoing DBS implantation for movement disorders. In addition to standard-of-care subcortical mapping using micro-electrode recording (MER) and macro-stimulation mapping during DBS placement, cortical local field potentials (LFPs) will be simultaneously recorded from primary motor (M1) and somatosensory (S1) cortical areas by placement of a temporary strip electrode (1X6) in the subdural space. Appropriate localization of this grid over M1 and S1 will be confirmed by the so-called phase-reversal of somatosensory evoked potentials (SSEPs). Once M1 is localized, the strip electrode over M1 will be used to produce motor evoked potentials to contralateral hand muscles from direct cortical stimulation (DCMEPs). The stimulation threshold of the DCMEPs will be used as a direct measure of the excitability of the cortical spinal tract and compared with and without stimulation of the VOP/VIM nuclei. Cortical and subcortical LFPs will be obtained alongside electromyographic (EMG) data while the patient performs contralateral upper extremity movement tasks measuring velocity, grip strength, and strength modulation and while the patient perform a variety of articulation exercises. Along with the DCMEP stimulation thresholds, these parameters of motor output will be obtained both with and without VOP/VIM stimulation to assess for stimulation induced potentiation of motor output.

ELIGIBILITY:
Inclusion Criteria:

* Essential tremor patients who are scheduled to undergo deep brain stimulation surgery at UPMC Presbyterian with asymmetric essential tremor symptoms will be included, with the tested limb corresponding to the least affected arm to better approximate normal function. These patients are implanted bilaterally regardless of symptom laterality, as the natural history of essential tremor indicates eventual bilateral symptoms.
* Parkinson's Disease patients who are scheduled to undergo deep brain stimulation surgery at UPMC Presbyterian with a history of Parkinson's Disease will also be recruited for intra-operative stimulation of their STN-targeted implants, to assess if VIM/VOP has high specificity for improving motor output.

Confirmation that subjects' terms of insurance coverage for their standard of care procedure will not be altered by study enrollment.

Exclusion Criteria:

* Patients will be excluded from the study if there is any seizure history, to avoid the increased epileptogenic risk of intraoperative stimulation.
* Patients with significant bilateral tremor that precludes completion of motor tasks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Electromyography Activity | 14 days
  The investigators will record electromyography activity (EMG) to measure the motor evoked potentials of upper limb and facial muscles. At the end of the procedures these needles and/or the superficial adhesive electrodes will be removed. Based on the preliminary data, the investigators will consider the number of participants with at least an 18% increase in muscle activation as minimally acceptable.

SECONDARY OUTCOMES:
Facial Muscle Motor Function - Muscle Strength | 14 days
  The investigators will use electromyography (EMG) testing to measure muscle strength produced by the subject during isometric facial movements (e.g. smile, tongue out, puckered lips, and open-close mouth). Amplitude of movement will be calculated by Area-Under-the-Curve with units of uV^2/ms. Based on the preliminary data, the investigators will consider the number of participants with an increase of 50% in ROM as a minimally acceptable improvement in muscle strength.
Facial Muscle Motor Function - Range of Motion | 14 days
  The investigators will use electromyography (EMG) testing to measure range of motion produced by the subject during isometric facial movements (e.g. smile, tongue out, puckered lips, and open-close mouth). Based on the preliminary data, the investigators will consider the number of participants with an increase of 50% in ROM as a minimally acceptable improvement.
Speech Intelligibility | 14 days
  The investigators will use the Assessment of Intelligibility of Dysarthric Speech (AIDS) to assess the quality of communication and intelligibility of speech at both word- and sentence-level. Intelligibility is calculated as the percentage of words correctly identified in the single-word task, and as the percentage of correctly transcribed words and speech rate (in words per minute) in the sentence task. Based on the preliminary data, the investigators will consider the number of participants with an improvement of 5% correctly transcribed to be minimally acceptable.
Dexterity of Articulation AMRs | 14 days
  The investigators will measure dexterity of articulation by alternating motion rates (AMRs) of the repetitive plosive sound (pah, tah, and kah). Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.
Dexterity of Articulation SMRs | 14 days
  The investigators will measure dexterity of articulation by sequential motion rates (SMRs) of the repetitive plosive sound (pah, tah, and kah). Based on the preliminary data, the investigators will consider the number of participants with an improvement of 10% in the rate to be minimally acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gonzalez-Martinez, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, may be shared with other researchers for the purpose of data analysis and collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of the trial upon publication of the first manuscript. Estimation is 7 years from enrollment of the first participant.
Access Criteria: Data must be directly requested from the PI and will be shared upon completion of the necessary data-sharing agreement to protect confidential patient information.